CLINICAL TRIAL: NCT03124069
Title: A Development Study to Evaluate a Nasal Mask for the Treatment of Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIA-211
Record Dates: First submitted 2017-04-11; First posted 2017-04-21 (Actual); Results first posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-06

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: After a period of baseline, all enrolled participants will be put on the same trial mask.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- F&P Saturn (Experimental): Participants will be placed on this arm for a total of 14 ± 5 days from Visit 2. Participants will be using the trial nasal mask during this treatment arm.
  Interventions: Device: F&P Saturn

INTERVENTIONS:
Device: F&P Saturn — Participants will be placed on this arm for a total of 14 ± 5 days from Visit 2. Participants will be using the trial nasal mask during this treatment arm.

SUMMARY:
This investigation is designed to evaluate the comfort, ease of use and performance of a trial nasal mask for the treatment of Obstructive Sleep Apnea (OSA) in the home environment.

DETAILED DESCRIPTION:
The investigation is a prospective, non-randomized, non-blinded study. Up to 45 OSA patients who currently use a nasal or nasal pillows mask will be recruited

This study will involve a baseline (Visit One) data gathering with the participant's PAP therapy and their usual mask. This will be followed by the participants being fitted with the trial nasal mask for use in-home (Visit Two). The participant then will come in to return the mask (Visit Three) and give feedback on their experience using the mask in home in the form of a structured interview during Visit Three. The maximum amount of time the participants will be exposed to the trial mask in-home will be 14 ± 5 days from Visit Two.

The mask and CPAP (if used from the loan research pool) will be returned to the institution at the conclusion of the trial and participant will return to their usual mask and therapy device for the treatment of Obstructive Sleep Apnea.

Neither the investigators nor the participants will be blinded to the study.

ELIGIBILITY:
Inclusion Criteria:

* AHI ≥ 5 from diagnostic PSG night
* Aged 22 and over (FDA defined as adult)
* Either prescribed APAP, CPAP or Bi-Level PAP for OSA
* Existing nasal or nasal pillows mask users (preferable 70%:30% split)
* Fluent in spoken and written English

Exclusion Criteria:

* Inability to give informed consent
* Patient intolerant to CPAP therapy
* Anatomical or physiological conditions making PAP therapy inappropriate
* Current diagnosis of respiratory disease or CO2 retention
* Pregnant or think they may be pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2017-05-26 (Actual); Study Completion 2017-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trials of Florida, South Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared with any other researchers or parties.

RESULTS

PARTICIPANT FLOW:
Groups:
- F&P Nasal Mask: Participants will be placed on this arm for a total of 14 ± 5 days from Visit 2. Participants will be using the trial nasal mask during this treatment arm.
Period: Overall Study
Arm/Group | F&P Nasal Mask
Started | 37
Completed | 37
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- F&P Nasal: Participants will be placed on this arm for a total of 14 ± 5 days from Visit 2. Participants will be using the trial nasal mask during this treatment arm.
Arm/Group | F&P Nasal
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 37
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Comfort Compared to Their Usual Mask.
Description: Comfort reported from participants questionnaires to evaluate the use of the F&P nasal mask for treatment of Obstructive Sleep Apnea
Time Frame: 14 ± 5 days In-Home
Measure: Count of Participants; unit: Participants
Groups:
- F&P Nasal: Participants will be placed on this arm for a total of 14 ± 5 days from Visit 2. Participants will be using the trial nasal mask during this treatment arm.
  .
Arm/Group | F&P Nasal
Number analyzed (Participants) | 37
Participants
  Much better | 17
  Better | 4
  Same | 9
  Worse | 6
  Much Worse | 1

2. Primary Outcome: Number of Participants PAP Device Performance Reporting
Description: Determined from data recorded from the PAP device to evaluate the use of the F&P nasal mask for treatment of Obstructive Sleep Apnea
Time Frame: 14 ± 5 days In-Home
Measure: Count of Participants; unit: Participants
Arm/Group | F&P Nasal
Number analyzed (Participants) | 37
Participants
  Better than usual mask | 9
  Same as usual mask | 13
  Worse than usual mask | 2
  No data | 13

3. Primary Outcome: Number of Participants Subjective Performance Rating of the Nasal Mask
Description: Performance reported from participants questionnaires to evaluate the use of the F&P nasal mask for treatment of Obstructive Sleep Apnea
Time Frame: 14 ± 5 days In-Home
Measure: Count of Participants; unit: Participants
Arm/Group | F&P Nasal
Number analyzed (Participants) | 37
Participants
  Very good | 23
  Good | 6
  Acceptable | 4
  Poor | 4
  Very Poor | 0

4. Primary Outcome: Number of Participants Subjective Reporting of Nasal Mask Usability
Description: Usability reported from participants questionnaires to evaluate the use of the F&P nasal mask for treatment of Obstructive Sleep Apnea
Time Frame: During Visit Two - 20 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | F&P Nasal
Number analyzed (Participants) | 37
Participants
  Very Easy | 23
  Easy | 9
  Acceptable | 5
  Difficult | 0
  Very Difficult | 0

5. Primary Outcome: Number of Participants Subjective Recording of Ease of Nasal Mask Use.
Description: Ease of use reported from participants questionnaires to evaluate the use of the F&P nasal mask for treatment of Obstructive Sleep Apnea
Time Frame: 14 ± 5 days In-Home
Measure: Count of Participants; unit: Participants
Arm/Group | F&P Nasal Mask
Number analyzed (Participants) | 37
Participants
  Very Easy | 23
  Easy | 9
  Acceptable | 5
  Difficult | 0
  Very Difficult | 0

6. Secondary Outcome: Number of Participants Leak Compared to Usual Mask
Description: Leak data recorded from PAP device to evaluate the use of the F&P nasal mask for treatment of Obstructive Sleep Apnea
Time Frame: 14 ± 5 days In-Home
Measure: Count of Participants; unit: Participants
Arm/Group | F&P Nasal
Number analyzed (Participants) | 37
Participants
  No Data | 13
  Better than current mask | 9
  Same as current mask | 13
  Worse than current mask | 2

7. Secondary Outcome: Number of Participants With Correct Nasal Mask Size Determination
Description: Sizing determined from a customized fitting tool to evaluate the use of the F&P nasal mask for treatment of Obstructive Sleep Apnea
Time Frame: 1 day-time appointment (1 hour)
Measure: Count of Participants; unit: Participants
Arm/Group | F&P Nasal Mask
Number analyzed (Participants) | 37
Participants
  Correct | 22
  In between sizes | 6
  Incorrect | 9

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | F&P Nasal Mask
All-Cause Mortality (participants affected / at risk) | 0/37
Serious Adverse Events (participants affected / at risk) | 0/37
Other Adverse Events (participants affected / at risk) | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-12): https://cdn.clinicaltrials.gov/large-docs/69/NCT03124069/Prot_SAP_002.pdf